CLINICAL TRIAL: NCT02878291
Title: A Single-center, Open, Phase I Clinical Trial to Evaluate Safety of Meningococcal ACYW135 Polysaccharide Conjugate Vaccine in Healthy Volunteers Aged Above 3 Months
Brief Title: Safety Study of Meningococcal ACYW135 Polysaccharide Conjugate Vaccine in Healthy Volunteers Aged Above 3 Months
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Collaborators: Guangxi Center for Disease Control and Prevention (Other Government); Sanjiang Center for Disease Control and Prevention (Unknown); National Institutes for Food and Drug Control, China (Other); Air Force Military Medical University, China (Other); Simoon Record Pharma Information Consulting Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201518603
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Meningitis, Meningococcal
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High dose Group (Experimental): Received Vaccine: Meningococcal ACYW135 Polysaccharide Conjugate Vaccine,40μg/dose
  Interventions: Biological: Meningococcal ACYW135 Polysaccharide Conjugate Vaccine
- low dose Group (Experimental): Received Vaccine: Meningococcal ACYW135 Polysaccharide Conjugate Vaccine,20μg/dose
  Interventions: Biological: Meningococcal ACYW135 Polysaccharide Conjugate Vaccine

INTERVENTIONS:
Biological: Meningococcal ACYW135 Polysaccharide Conjugate Vaccine — Group 1:3/2/1 dose(s) according to age of subjects. Single intramuscular dose contains 10 µg each of Serogroup A, C, Y, and W135 polysaccharide conjugated to Tetanus Toxoids.
  Other Names: Menwaycon
  Arms: High dose Group
Biological: Meningococcal ACYW135 Polysaccharide Conjugate Vaccine — Group 2:3/2/1 dose(s) according to age of subjects. Single intramuscular dose contains 5 µg each of Serogroup A, C, Y, and W135 polysaccharide conjugated to Tetanus Toxoids.
  Other Names: Menwaycon
  Arms: low dose Group

SUMMARY:
The purpose of this study is to evaluate safety of meningococcal ACYW135 polysaccharide conjugate vaccine in healthy volunteers aged above 3 Months

ELIGIBILITY:
Inclusion Criteria:

* 3-11 months health infants who haven't immuned with Meningococcal A and C Conjugate Vaccine and population above 1 year old who have't given boost immunity.
* Subject or legal representative who consent and has signed written informed consent.
* Subject who did't immune with any live vaccine within 14 days and inactivated vaccine within 7 days before vaccination.
* Subject and parent/guardian who is able to comply with all study procedures.
* Axillary temperature ≤37.0 ℃.

Exclusion Criteria:

* History of allergy，eclampsia, epilepsy, encephalopathy and mental disease or family disease.
* Allergic history after vaccination.
* History of meningitis infection disease.
* Acute Febrile illness and Infectious Diseases.
* Febrile illness (temperature ≥ 38°C) in the 3 days.
* Immunodeficiency diseases patients who administered with immunosuppressive agents.
* Children within 1 year old with abnormal labor, asphyxia rescue history,congenital malformations,genetic defects, eccyliosis or severe chronic disease.
* Liver and kidney or cardiopulmonary disease，acute hypertension and diabetes.
* In pregnancy or lactation or pregnant women.
* Subject who plan to participate in or is in any other drug clinical trial.
* Meningococcal vaccine contraindication.
* Any condition that, in the judgment of investigator, may affect trial assessment.

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events during a 30 day follow-up period after each vaccination | 30 day after each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Du lin, Master, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (1):
- Sanjiang Center for Disease Control and Prevention, Sanjiang, Guangxi, China

IPD SHARING:
Plan to Share IPD: No